CLINICAL TRIAL: NCT07386366
Title: Evaluation of Soft Tissue Healing and Antibacterial Effectiveness of Triclosan-Coated Polyglactin 910 Sutures After Impacted Mandibular Third Molar Surgery: A Randomized Double-Blind Split-Mouth Clinical Trial
Brief Title: Wound Healing and Bacterial Adherence With Triclosan-Coated Sutures After Mandibular Impacted Third Molar Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Le Khanh Huyen Nguyen, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3774/ĐHYD-HĐĐĐ
Record Dates: First submitted 2026-01-19; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Impacted Mandibular Third Molar; Postoperative Wound Healing
Keywords: Triclosan-coated suture; Polyglactin 910; Impacted third molar surgery; Mandibular third molar; Oral surgery; Postoperative wound healing; Bacterial adhesion; Antibacterial suture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Triclosan-coated → Non-coated (Other): Two-period crossover. Period 1 (first surgery): triclosan-coated polyglactin 910 suture. Period 2 (second surgery, approximately 4 weeks later): non-coated polyglactin 910 suture. Operated side (right/left) may vary by case; assignment is based on surgery order.
  Interventions: Device: Triclosan-coated Polyglactin 910 suture; Device: Non-coated polyglactin 910 suture
- Sequence 2: Non-coated → Triclosan-coated (Other): Two-period crossover. Period 1 (first surgery): non-coated polyglactin 910 suture. Period 2 (second surgery, approximately 4 weeks later): triclosan-coated polyglactin 910 suture. Operated side (right/left) may vary by case; assignment is based on surgery order.
  Interventions: Device: Triclosan-coated Polyglactin 910 suture; Device: Non-coated polyglactin 910 suture

INTERVENTIONS:
Device: Triclosan-coated Polyglactin 910 suture — Absorbable braided polyglactin 910 suture coated with triclosan for wound closure after mandibular impacted third molar surgery.
Device: Non-coated polyglactin 910 suture — Absorbable braided polyglactin 910 suture without triclosan coating for wound closure after mandibular impacted third molar surgery.

SUMMARY:
The goal of this clinical trial is to learn if triclosan-coated absorbable stitches (polyglactin 910 sutures coated with triclosan, an antibacterial agent) help soft tissue heal better and have fewer bacteria stuck to the stitches after lower impacted wisdom tooth surgery in adults aged 18 to 35 years.

The main questions it aims to answer are:

1. Does triclosan-coated polyglactin 910 suture lead to better soft-tissue wound healing than non-coated polyglactin 910 suture on postoperative days 3, 5, and 7 after mandibular impacted third molar surgery?
2. Does triclosan-coated polyglactin 910 suture result in a lower oral bacterial load adhered to the suture material than non-coated polyglactin 910 suture on postoperative days 3, 5, and 7 after mandibular impacted third molar surgery?

Participants will:

* Have surgery to remove two similar lower impacted wisdom teeth (one on each side)
* Receive triclosan-coated stitches on one side and standard stitches on the other side, with the side assignment chosen at random
* Return for follow-up visits on day three, day five, and day seven after surgery for healing checks, simple ratings of pain and swelling, and collection of a small stitch sample for bacterial testing.

DETAILED DESCRIPTION:
This randomized, double-blind, two-period crossover clinical trial evaluates the antibacterial performance of triclosan-coated polyglactin 910 sutures compared with standard (non-coated) polyglactin 910 sutures following impacted mandibular third molar surgery. The study is designed to determine whether triclosan coating reduces bacterial adherence/amount on suture material during early postoperative healing and to examine associated soft-tissue healing.

Each participant undergoes two separate surgical extractions of impacted mandibular third molars performed on different occasions 4 weeks apart. The operated side (right or left) may vary by case and is recorded; treatment assignment is based on surgery order (period 1 versus period 2). Participants are randomized to one of two sequences: (A) triclosan-coated suture in the first surgery followed by non-coated suture in the second surgery, or (B) the reverse sequence. Standardized perioperative management is used across both periods to reduce procedural variability.

Masking is maintained for participants and outcome assessors. Allocation is concealed and documented for analysis after data collection. For each surgery, follow-up assessments are conducted during the first postoperative week using prespecified clinical evaluations and laboratory testing of a small collected suture segment, with consistent follow-up timing across both periods. Follow-up visits occur on postoperative days 3, 5, and 7 after each surgery.

The crossover design enables within-participant comparisons between suture types, reducing inter-individual variation in oral microbiota and healing response. The 4-week interval between procedures is intended to minimize carryover effects from the first surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 35 years.
* American Society of Anesthesiologists (ASA) physical status I or II.
* Presence of two symmetric impacted mandibular third molars with the same level of difficulty according to the Pell-Gregory and Winter classification; the difference in angulation between the two third molars is no more than 15 degrees.
* No use of topical or systemic antibiotics for at least 4 weeks before surgery.
* Able and willing to provide written informed consent.
* No active infection associated with the mandibular third molar at the time of enrollment.

Exclusion Criteria:

* Pregnant or breastfeeding.
* Allergy to local anesthetic (2% lidocaine with 1:100,000 epinephrine) or any medications used in the study.
* Radiographic findings suggestive of a tumor or cyst associated with the impacted mandibular third molar.
* Participant withdraws consent or does not agree to continue participation.
* Unable to attend scheduled follow-up visits.
* Difference in surgical extraction time between the two procedures is 12 minutes or more.
* Suture loss/loosening before completion of the final assessment time point.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Oral bacterial load on suture material (real-time PCR) | Postoperative days 3, 5, and 7 after each surgery (period 1 and period 2).
  Bacterial load on collected suture segments quantified using real-time polymerase chain reaction (real-time PCR) and compared between triclosan-coated and non-coated polyglactin 910 sutures within participants in a two-period crossover design.

SECONDARY OUTCOMES:
Soft-tissue wound healing (IPR score) | Postoperative days 3, 5, and 7 after each surgery (Period 1 and Period 2).
  Soft-tissue healing will be assessed using the Inflammatory-Proliferative-Remodeling (IPR) Wound Healing Score (Hamzani 2018). The total IPR score ranges from 0 to 8, with higher scores indicating better healing. At each visit, eight parameters are scored as 0 (unfavorable) or 1 (favorable): bleeding (spontaneous or on palpation), granulation tissue, hematoma, tissue color, incision margins, suppuration, edema (VAS 0-100 mm; 0 = 51-100 mm, 1 = 0-50 mm), and pain (VAS 0-100 mm; 0 = 51-100 mm, 1 = 0-50 mm).
Postoperative pain (VAS 0-100) | Postoperative days 3, 5, and 7 after each surgery (period 1 and period 2).
  Participant-reported pain measured on a 0-100 visual analog scale (VAS), where 0 indicates no pain and 100 indicates the worst imaginable pain.
Postoperative swelling (VAS 0-100) | Postoperative days 3, 5, and 7 after each surgery (period 1 and period 2).
  Participant-reported swelling measured on a 0-100 visual analog scale (VAS), where 0 indicates no swelling and 100 indicates the worst imaginable swelling.

CONTACTS AND LOCATIONS:
Overall Officials: Son Hoang Le, Study Chair — Department of Oral Surgery, Faculty of Dentistry, University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- Specialized Dental Clinic, University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes